CLINICAL TRIAL: NCT05163743
Title: COVID-19 Vaccination in Subjects With Obesity: Impact of Metabolic Health and the Role of a Ketogenic Diet
Brief Title: Diet and COVID-19 Vaccination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Lucio Gnessi, Principal Investigator, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KDC19090421
Record Dates: First submitted 2021-12-16; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Obesity
Keywords: Ketogenic Diet, COVID-19, VAT, Obesity
MeSH Terms: conditions — Obesity; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet-obese (Experimental): LCKD (1200-1400kcal/day) low in carbohydrates (<50g per day) with a moderate protein intake (1-1.5g/kg of ideal body mass) but otherwise no other dietary restrictions. The participants will be counselled by a trained nutritionist at baseline and every two weeks, and compliance will be assessed through a 3-day dietary recall at each follow up visit and capillary beta hydroxybutyrate levels as well as urinary acetoacetate levels. The follow up visits take place at the time of the first vaccine dose, two weeks after the first vaccine dose, one week after the second vaccine dose. Then, gradual reintroduction of carbohydrates will take place following the second vaccine dose.
  Interventions: Dietary Supplement: Low Calorie Ketogenic Diet

INTERVENTIONS:
Dietary Supplement: Low Calorie Ketogenic Diet — The very low-carbohydrate diet will be hypo caloric and aim to provide less than 50 g of carbohydrates per day. the participants will be counseled to choose vegetarian and healthy sources of fat and protein and to avoid trans fat. Then, gradual reintroduction of carbohydrates will take place following the second vaccine dose.

SUMMARY:
Recently, obesity and excess visceral fat were shown to be major risk factors for the development of complications following Covid 19 infection. Recently, KDs have been suggested as possible weapons to tame the cytokine storm being described in those developing complications upon COVID-19 infection, and preclinical evidence strongly supports the hypothesis, with mouse models of COVID-19 infection in the elderly reporting strikingly better outcomes upon consumption of a KD. Short-term interventions that use low-calorie ketogenic diets may be prescribed for selected overweight or obese patients with type 2 diabetes or prediabetes.

No data is available on the impact of a ketogenic diet on immune modulation following vaccination. We herein aim at investigating whether obesity and unhealthy body composition are associated with poor seroconversion following the upcoming COVID-19 vaccine administration, and whether consumption of a KD before and between COVID-19 vaccine doses leads to better immune response in obese subjects. 24 obese patients will be assigned to follow a LCKD regimen for 5 weeks.

DETAILED DESCRIPTION:
Recently, obesity and excess visceral fat were shown to be major risk factors for the development of complications following Covid 19 infection. Recently, KDs have been suggested as possible weapons to tame the cytokine storm being described in those developing complications upon COVID-19 infection, and preclinical evidence strongly supports the hypothesis, with mouse models of COVID-19 infection in the elderly reporting strikingly better outcomes upon consumption of a KD. Short-term interventions that use low-calorie ketogenic diets may be prescribed for selected overweight or obese patients with type 2 diabetes or prediabetes.

No data is available on the impact of a ketogenic diet on immune modulation following vaccination. We herein aim at investigating whether obesity and unhealthy body composition are associated with poor seroconversion following the upcoming COVID-19 vaccine administration, and whether consumption of a KD before and between COVID-19 vaccine doses leads to better immune response in obese subjects. 24 patients will be assigned to follow a low-calorie ketogenic diet (LCKD). Outcome measures will be antiSARS-CoV-2 antibodies, cell mediated response to SARS CoV-2, anthropometric parameters, vital signs, metabolic profile, and body composition. The patients will be assessed at baseline (T0) and every two weeks (T1, T2) as they receive both SARS Cov-2 vaccination doses up to 1 week after the second dose (T3) when they will be finally evaluated and carbohydrate reintroduction takes place. Patients will be given support and counselling to enhance their compliance. Anthropometric parameters such as body weight, blood pressure (systolic and diastolic), heart rate, waist and hip circumference will be measured at baseline (T0), every two weeks up to the end of the trial (T3).

Blood and urine chemistry Complete Blood Count (CBC), electrolytes (chloride, calcium, potassium, sodium, magnesium), fasting glucose, insulin, lipids (total and fractionated cholesterol and triglycerides) and proteins, C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR), plasma creatinine, blood urea nitrogen (BUN), alanine transferase (AST), aspartate transaminase (ALT), uric acid, beta hydroxy butyrate and estimated Glomerular Filtration Rate (using the Modification of Diet in Renal Disease study equation MDRD-eGFR) will be determined

AntiSARS-CoV-2 antibodies: antibodies will be quantified by enzyme-linked immunosorbent assay using the appropriate antigen at T3 and T4 in all arms. The cell mediated response to SARS CoV-2 will be analyzed by taking whole blood that will be stimulated with immune ligands.

Data obtained will be expressed as mean values ±Standard Deviation (SD) and finally processed to ascertain whether statistical differences among them can be demonstrated, using appropriate methods. In particular, the analysis of variance (ANOVA) at different times will be used for efficacy and safety data, such as weight reduction, changes in anthropometric measures, and variation of the metabolic parameters. P values <0.05 will be considered statistically significant.

ELIGIBILITY:
* BMI ≥35.0 kg/m2 with comorbidities or BMI≥40
* Stable body weight (less than 5 kg self-reported change during the previous 3 months)
* Informed consent obtained before any trial-related activity takes place Exclusion criteria
* Stage 3-5 CKD (GFR<60 ml/min)
* Type 1 diabetes
* Uncontrolled type 2 diabetes
* Previous infection with SARS CoV-2
* Immunodeficiency or immunomodulating treatment
* Treatment with anti-obesity medications or other medications potentially affecting body weight or SGLT2 inhibitors
* Pregnancy and lactation
* Previous gout episodes
* Cardio and cerebrovascular accidents in the preceding 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-23 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
AntiSARS-CoV-2 antibodies | 5 weeks
  antibodies will be quantified by enzyme-linked immunosorbent assay at week 0 and 5
Cell mediated response to SARS CoV-2 | 5 weeks
  whole blood will be stimulated with immune ligands within 8 h from blood collection.

SECONDARY OUTCOMES:
Body weight | 5 weeks
  Body weight will be obtained with the subjects wearing very light clothing and no shoes, and with an empty bladder. The same scale will be used throughout the study. The scale will be calibrated.
Waist Circumference | 5 weeks
  Waist circumference will be measured on subjects while semi clothed, standing with their feet close together and their weight equally distributed on each leg. Subjects will be asked to breath normally. Circumference will be taken at the midpoint between the lower rib margin and the iliac crest.
Triglycerides, glucose, insulin, ESR, CRP, ferritin | 5 weeks
  All biochemical parameters will be measured according to local laboratory standards.

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Gnessi, MD PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe M, Risi R, De Giorgi F, Tuccinardi D, Mariani S, Basciani S, Lubrano C, Lenzi A, Gnessi L. Obesity treatment within the Italian national healthcare system tertiary care centers: what can we learn? Eat Weight Disord. 2021 Apr;26(3):771-778. doi: 10.1007/s40519-020-00936-1. Epub 2020 May 25. PMID 32451949
- [Background] Mariani S, Fiore D, Varone L, Basciani S, Persichetti A, Watanabe M, Saponara M, Spera G, Moretti C, Gnessi L. Obstructive sleep apnea and bone mineral density in obese patients. Diabetes Metab Syndr Obes. 2012;5:395-401. doi: 10.2147/DMSO.S37761. Epub 2012 Nov 7. PMID 23152692
- [Background] Lonardo A, Mantovani A, Lugari S, Targher G. Epidemiology and pathophysiology of the association between NAFLD and metabolically healthy or metabolically unhealthy obesity. Ann Hepatol. 2020 Jul-Aug;19(4):359-366. doi: 10.1016/j.aohep.2020.03.001. Epub 2020 Mar 21. PMID 32349939
- [Background] Dwivedi AK, Dubey P, Cistola DP, Reddy SY. Association Between Obesity and Cardiovascular Outcomes: Updated Evidence from Meta-analysis Studies. Curr Cardiol Rep. 2020 Mar 12;22(4):25. doi: 10.1007/s11886-020-1273-y. PMID 32166448
- [Background] Okamura T, Hashimoto Y, Hamaguchi M, Obora A, Kojima T, Fukui M. Ectopic fat obesity presents the greatest risk for incident type 2 diabetes: a population-based longitudinal study. Int J Obes (Lond). 2019 Jan;43(1):139-148. doi: 10.1038/s41366-018-0076-3. Epub 2018 May 1. PMID 29717276
- [Background] Palermo A, Tuccinardi D, Defeudis G, Watanabe M, D'Onofrio L, Lauria Pantano A, Napoli N, Pozzilli P, Manfrini S. BMI and BMD: The Potential Interplay between Obesity and Bone Fragility. Int J Environ Res Public Health. 2016 May 28;13(6):544. doi: 10.3390/ijerph13060544. PMID 27240395
- [Background] Arboleda S, Vargas M, Losada S, Pinto A. Review of obesity and periodontitis: an epidemiological view. Br Dent J. 2019 Aug;227(3):235-239. doi: 10.1038/s41415-019-0611-1. PMID 31399683
- [Background] Watanabe M, Caruso D, Tuccinardi D, Risi R, Zerunian M, Polici M, Pucciarelli F, Tarallo M, Strigari L, Manfrini S, Mariani S, Basciani S, Lubrano C, Laghi A, Gnessi L. Visceral fat shows the strongest association with the need of intensive care in patients with COVID-19. Metabolism. 2020 Oct;111:154319. doi: 10.1016/j.metabol.2020.154319. Epub 2020 Jul 23. PMID 32712222
- [Background] Petrilli CM, Jones SA, Yang J, Rajagopalan H, O'Donnell L, Chernyak Y, Tobin KA, Cerfolio RJ, Francois F, Horwitz LI. Factors associated with hospital admission and critical illness among 5279 people with coronavirus disease 2019 in New York City: prospective cohort study. BMJ. 2020 May 22;369:m1966. doi: 10.1136/bmj.m1966. PMID 32444366
- [Background] Watanabe M, Risi R, Tuccinardi D, Baquero CJ, Manfrini S, Gnessi L. Obesity and SARS-CoV-2: A population to safeguard. Diabetes Metab Res Rev. 2020 Oct;36(7):e3325. doi: 10.1002/dmrr.3325. Epub 2020 Jun 11. PMID 32314503
- [Background] McLarnon A. Obesity: influenza immunity impaired in obesity. Nat Rev Endocrinol. 2011 Nov 15;8(1):3. doi: 10.1038/nrendo.2011.199. No abstract available. PMID 22083087
- [Background] Andersen CJ, Murphy KE, Fernandez ML. Impact of Obesity and Metabolic Syndrome on Immunity. Adv Nutr. 2016 Jan 15;7(1):66-75. doi: 10.3945/an.115.010207. Print 2016 Jan. PMID 26773015
- [Background] Painter SD, Ovsyannikova IG, Poland GA. The weight of obesity on the human immune response to vaccination. Vaccine. 2015 Aug 26;33(36):4422-9. doi: 10.1016/j.vaccine.2015.06.101. Epub 2015 Jul 8. PMID 26163925
- [Background] Neidich SD, Green WD, Rebeles J, Karlsson EA, Schultz-Cherry S, Noah TL, Chakladar S, Hudgens MG, Weir SS, Beck MA. Increased risk of influenza among vaccinated adults who are obese. Int J Obes (Lond). 2017 Sep;41(9):1324-1330. doi: 10.1038/ijo.2017.131. Epub 2017 Jun 6. PMID 28584297
- [Background] Gardner CD, Trepanowski JF, Del Gobbo LC, Hauser ME, Rigdon J, Ioannidis JPA, Desai M, King AC. Effect of Low-Fat vs Low-Carbohydrate Diet on 12-Month Weight Loss in Overweight Adults and the Association With Genotype Pattern or Insulin Secretion: The DIETFITS Randomized Clinical Trial. JAMA. 2018 Feb 20;319(7):667-679. doi: 10.1001/jama.2018.0245. PMID 29466592
- [Background] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428
- [Background] Vandanmagsar B, Youm YH, Ravussin A, Galgani JE, Stadler K, Mynatt RL, Ravussin E, Stephens JM, Dixit VD. The NLRP3 inflammasome instigates obesity-induced inflammation and insulin resistance. Nat Med. 2011 Feb;17(2):179-88. doi: 10.1038/nm.2279. Epub 2011 Jan 9. PMID 21217695
- [Background] Youm YH, Nguyen KY, Grant RW, Goldberg EL, Bodogai M, Kim D, D'Agostino D, Planavsky N, Lupfer C, Kanneganti TD, Kang S, Horvath TL, Fahmy TM, Crawford PA, Biragyn A, Alnemri E, Dixit VD. The ketone metabolite beta-hydroxybutyrate blocks NLRP3 inflammasome-mediated inflammatory disease. Nat Med. 2015 Mar;21(3):263-9. doi: 10.1038/nm.3804. Epub 2015 Feb 16. PMID 25686106
- [Background] Ang QY, Alexander M, Newman JC, Tian Y, Cai J, Upadhyay V, Turnbaugh JA, Verdin E, Hall KD, Leibel RL, Ravussin E, Rosenbaum M, Patterson AD, Turnbaugh PJ. Ketogenic Diets Alter the Gut Microbiome Resulting in Decreased Intestinal Th17 Cells. Cell. 2020 Jun 11;181(6):1263-1275.e16. doi: 10.1016/j.cell.2020.04.027. Epub 2020 May 20. PMID 32437658
- [Background] Choi IY, Piccio L, Childress P, Bollman B, Ghosh A, Brandhorst S, Suarez J, Michalsen A, Cross AH, Morgan TE, Wei M, Paul F, Bock M, Longo VD. A Diet Mimicking Fasting Promotes Regeneration and Reduces Autoimmunity and Multiple Sclerosis Symptoms. Cell Rep. 2016 Jun 7;15(10):2136-2146. doi: 10.1016/j.celrep.2016.05.009. Epub 2016 May 26. PMID 27239035
- [Background] Yasuda K, Takeuchi Y, Hirota K. The pathogenicity of Th17 cells in autoimmune diseases. Semin Immunopathol. 2019 May;41(3):283-297. doi: 10.1007/s00281-019-00733-8. Epub 2019 Mar 19. PMID 30891627
- [Background] Sukkar SG, Bassetti M. Induction of ketosis as a potential therapeutic option to limit hyperglycemia and prevent cytokine storm in COVID-19. Nutrition. 2020 Nov-Dec;79-80:110967. doi: 10.1016/j.nut.2020.110967. Epub 2020 Aug 10. PMID 32942131
- [Background] Bradshaw PC, Seeds WA, Miller AC, Mahajan VR, Curtis WM. COVID-19: Proposing a Ketone-Based Metabolic Therapy as a Treatment to Blunt the Cytokine Storm. Oxid Med Cell Longev. 2020 Sep 9;2020:6401341. doi: 10.1155/2020/6401341. eCollection 2020. PMID 33014275
- [Background] Ryu S, Shchukina I, Youm YH, Qing H, Hilliard BK, Dlugos T, Zhang X, Yasumoto Y, Booth CJ, Fernandez-Hernando C, Suarez Y, Khanna KM, Horvath TL, Dietrich MO, Artyomov MN, Wang A, Dixit VD. Ketogenesis restrains aging-induced exacerbation of COVID in a mouse model. bioRxiv [Preprint]. 2020 Sep 12:2020.09.11.294363. doi: 10.1101/2020.09.11.294363. PMID 33236006
- See also: Obesity and Overweight Factsheet June 2016 [08/04/2017]. — http://www.who.int/mediacentre/factsheets/fs311/en/